CLINICAL TRIAL: NCT02370095
Title: Treprostinil Sodium Inhalation for Patients At High Risk for ARDS: Effect on Oxygenation and Disease-related Biomarkers
Brief Title: Treprostinil Sodium Inhalation for Patients At High Risk for ARDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14-0490
Record Dates: First submitted 2015-01-30; First posted 2015-02-24 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: ARDS; Acute Lung Injury; Acute Respiratory Failure
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treprostinil inhalation solution (Active Comparator): Treprostinil will be randomized 2:1 to placebo. Treprostinil (6 mcg per breath) will be administered every 4 hours. The dose will increase from 6 to12 breaths (maximum 72 mcg) over the first 20 hours, maintained for 7 days, and tapered down over 3 days.
  Interventions: Drug: Treprostinil Inhalation Solution
- Placebo (Placebo Comparator): Placebo administration will be administered as above for the active arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treprostinil Inhalation Solution — Treprostinil inhalation solution administered as blinded marketed product
  Other Names: TYVASO
  Arms: Treprostinil inhalation solution
Drug: Placebo — Supplied by the manufacturer and similar to the active drug but containing no Treprostinil
  Other Names: Sterile saline solution
  Arms: Placebo

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is a rapidly progressing lung disease caused by a number of factors including pneumonia, sepsis and acute trauma that leads to reduced lung function and breathlessness. There are no pharmacological treatments approved for the treatment of ARDS. This pilot trial will study the safety and efficacy of Treprostinil sodium by inhalation for preventing the progression of acute hypoxemic respiratory failure to positive pressure ventilation and/or ARDS in patients at high risk.

DETAILED DESCRIPTION:
ARDS is defined by acute hypoxemia, respiratory failure and the presence of bilateral lung infiltrates. ARDS is a syndrome of inflammation and increased permeability that may coexist with left atrial or pulmonary capillary hypertension. Several recent trials in ARDS / ALI (Acute Lung Injury) have generated interest in the use of Prostacyclin (PGI2) and prostacyclin analogs in improving oxygenation in ARDS / ALI. PGI2 is an arachidonic acid metabolite naturally produced in the lung by endothelial cells, dendritic cells, smooth muscle cells and fibroblasts. PGI2 is a potent selective pulmonary vasodilator and inhibitor of platelet aggregation. The cellular effects include smooth muscle relaxation, inhibition of cell migration, decreased dextran permeability in epithelial cell cultures in vitro, decreased high tidal volume mechanical ventilation injury in mice and inhibition of fibroblast adhesion and differentiation. PGI2 has broad anti-inflammatory activity, inhibiting the production of Tumor necrosis factor alpha (TNFα), interleukin 1 beta (IL-1β), interleukin 6 (IL-6) and granulocyte macrophage colony-stimulating factor (GMCSF) in human alveolar macrophages.

The study objectives are:

1. To assess the feasibility of a randomized trial of treprostinil inhalation in patients with acute hypoxemic respiratory failure not requiring positive pressure ventilation.
2. To evaluate the tolerability of inhaled treprostinil for patients with acute hypoxemic respiratory failure
3. To assess the effect of treprostinil inhalation on oxygenation in patients with acute hypoxic respiratory failure with, or at risk for, development of ARDS
4. To assess the effect of treprostinil inhalation on various biomarkers thought to be related to the pathogenesis and/or clinical course of ARDS.

The hypothesis is: Treprostinil solution for inhalation (TYVASO) is safe and will improve oxygenation and other secondary outcomes related to acute hypoxemic respiratory failure and positive pressure ventilation initiation and duration, as well as exhibit effects on ARDS-related pro-inflammatory and pro-fibrotic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18-75 years.
2. Acute onset need for 4 liters per minute (LPM) or more of supplemental oxygen to maintain Arterial partial pressure of oxygen (PaO2) > 60 mmHg or arterial O2 saturation > 90% by pulse oximetry.
3. Acute unilateral pulmonary infiltrate/s on chest radiograph with no clinical evidence of left-sided heart failure. Bilateral infiltrates are acceptable as long as all other inclusion/exclusion criteria are met.

Exclusion Criteria:

1. No consent/inability to obtain consent
2. Presence of pulmonary embolism
3. Known diffuse alveolar hemorrhage from vasculitis
4. Known pre-existing severe obstructive or restrictive lung disease (FEV 1 < 40% predicted, total lung capacity (TLC) < 50 % predicted) or need for long-term supplemental oxygen therapy
5. Known significant left ventricular systolic dysfunction with left ventricular ejection fraction (LVEF) < 45% on echocardiogram.
6. Mean arterial pressure < 65 mmHg
7. Need for norepinephrine or dopamine dose > 12 mcg to maintain mean arterial pressure (MAP) > 65 mmHg
8. Severe chronic liver disease (Child-Pugh Score 11-15)
9. Moribund patient not expected to survive 24 hours
10. Corrected QT interval (QTc) interval > 500 ms on screening electrocardiogram
11. Pregnancy or breast feeding (Women of childbearing potential, defined as < 60 years of age, will require pregnancy testing.)
12. Burns > 40% total body surface
13. Acute Neurological Disease (that may impair the ability to ventilate without assistance)
14. Imminent need for intubation or non-invasive ventilation
15. Patient is Do Not Resuscitate/Do Not Intubate
16. Patient has a tracheotomy
17. Patient is currently receiving prostacyclin therapy [Epoprostenol (Flolan or Veletri), Iloprost (Ventavis), Treprostinil (Orenitram, oral) (Remodulin, IV or SC)]
18. Patient has a language barrier

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02; Primary Completion 2017-10-11 (Actual); Study Completion 2017-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert J Ford, MD, Principal Investigator — University of North Carolina, Chapel Hill; Shannon Carson, MD, Principal Investigator — University of North Carolina, Chapel Hill; Wayne H Anderson, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
only summary data via publication/abstract

REFERENCES:
- [Background] Zwissler B, Kemming G, Habler O, Kleen M, Merkel M, Haller M, Briegel J, Welte M, Peter K. Inhaled prostacyclin (PGI2) versus inhaled nitric oxide in adult respiratory distress syndrome. Am J Respir Crit Care Med. 1996 Dec;154(6 Pt 1):1671-7. doi: 10.1164/ajrccm.154.6.8970353.
- [Background] Walmrath D, Schneider T, Schermuly R, Olschewski H, Grimminger F, Seeger W. Direct comparison of inhaled nitric oxide and aerosolized prostacyclin in acute respiratory distress syndrome. Am J Respir Crit Care Med. 1996 Mar;153(3):991-6. doi: 10.1164/ajrccm.153.3.8630585.
- [Background] Walmrath D, Schneider T, Pilch J, Schermuly R, Grimminger F, Seeger W. Effects of aerosolized prostacyclin in severe pneumonia. Impact of fibrosis. Am J Respir Crit Care Med. 1995 Mar;151(3 Pt 1):724-30. doi: 10.1164/ajrccm.151.3.7881662.
- [Background] Domenighetti G, Stricker H, Waldispuehl B. Nebulized prostacyclin (PGI2) in acute respiratory distress syndrome: impact of primary (pulmonary injury) and secondary (extrapulmonary injury) disease on gas exchange response. Crit Care Med. 2001 Jan;29(1):57-62. doi: 10.1097/00003246-200101000-00015. PMID 11176161
- [Background] Dahlem P, van Aalderen WM, de Neef M, Dijkgraaf MG, Bos AP. Randomized controlled trial of aerosolized prostacyclin therapy in children with acute lung injury. Crit Care Med. 2004 Apr;32(4):1055-60. doi: 10.1097/01.ccm.0000120055.52377.bf. PMID 15071401
- [Background] Dorris SL, Peebles RS Jr. PGI2 as a regulator of inflammatory diseases. Mediators Inflamm. 2012;2012:926968. doi: 10.1155/2012/926968. Epub 2012 Jul 18. PMID 22851816
- [Background] Raychaudhuri B, Malur A, Bonfield TL, Abraham S, Schilz RJ, Farver CF, Kavuru MS, Arroliga AC, Thomassen MJ. The prostacyclin analogue treprostinil blocks NFkappaB nuclear translocation in human alveolar macrophages. J Biol Chem. 2002 Sep 6;277(36):33344-8. doi: 10.1074/jbc.M203567200. Epub 2002 Jun 24. PMID 12082102
- [Derived] Ford HJ, Anderson WH, Wendlandt B, Bice T, Ceppe A, Lanier J, Carson SS. Randomized, Placebo-controlled Trial of Inhaled Treprostinil for Patients at Risk for Acute Respiratory Distress Syndrome. Ann Am Thorac Soc. 2021 Apr;18(4):641-647. doi: 10.1513/AnnalsATS.202004-374OC. PMID 33095030

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was consented, randomized (Placebo) and baseline data was collected. However, before receiving treatment the subject deteriorated, and a protocol defined stopping rule was met. The subject was defined as completed. Baseline data were used in the analyses, and the AEs recorded are presented in the AE section.
Period: Overall Study
Arm/Group | Treprostinil Inhalation Solution | Placebo
Started | 10 | 4
Completed | 10 | 3
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who signed a consent are included in baseline measurements
Groups:
- Total: Total of all reporting groups
Arm/Group | Treprostinil Inhalation Solution | Placebo | Total
Number analyzed (Participants) | 10 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (13.1) | 51.8 (7.6) | 50.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8 | 3 | 11
  African-American | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in the Ratio of the Partial Pressure of Arterial Oxygen to the Fraction of Inspired Oxygen (PaO2/FiO2 Ratio)
Description: PaO2/FiO2 ratio
Time Frame: Change in PaO2/FiO2 ratio from day 0 to day 2.
Population: Determination of this endpoint was dependent on subject consent for collection of an arterial blood sample. A baseline measure was obtained from thirteen subjects. Samples were obtained from seven subjects at day 2, and two subjects at day 7 and none at day 28. Analysis was limited to change from baseline to day 2.
Measure: Mean (Standard Error); unit: P/F ratio
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 5 | 1
P/F ratio | 55.6 (31.2) | 161.1 (0)
Statistical Analysis 1: Comparison: Treprostinil Inhalation Solution vs Placebo; Only one placebo subject had data to allow for change from baseline to be calculated; Test type: Superiority; p = 0.2416, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in the Ratio of Peripheral Oxygen Saturation to Fraction of Inspired Oxygen (SaO2/FiO2)
Description: SaO2/FiO2
Time Frame: 0-12 days
Population: Intent to treat
Measure: Least Squares Mean (Standard Error); unit: S/F ratio
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 10 | 4
S/F ratio | 303.7 (22.0) | 382.3 (36.9)
Statistical Analysis 1: Comparison: Treprostinil Inhalation Solution vs Placebo; Test type: Superiority; p = 0.06, Mixed Models Analysis; The change in S/F ratio over time was evaluated using a mixed model for repeated measures

3. Secondary Outcome: Number of Days Not on a Ventilator
Description: Ventilator-free days
Time Frame: 0-28 days post enrollment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 10 | 4
days | 16.4 (14.1) | 28 (0)
Statistical Analysis 1: Comparison: Treprostinil Inhalation Solution vs Placebo; Test type: Superiority; p = 0.0679, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Subjects Who Required Bi-level Positive Airway Pressure (BiPAP) or Continuous Positive Airway Pressure (CPAP) Via Face Mask
Description: BiPAP / CPAP
Time Frame: 0-28 days
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 10 | 4
Participants | 2 | 1

5. Secondary Outcome: Acute Respiratory Distress Syndrome (ARDS) Associated Biomarkers
Description: Change in ARDS associated plasma biomarkers
Time Frame: Change from day 0 on days 3 and 7
Population: Too few samples were collected at the designated days 3 and 7 to provide informative data. Plasma samples were not analyzed.
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in the Central Venous Oxygen Saturation (SCVO2).
Description: SCVO2
Time Frame: Change in SCVO2 from Day 0 to 3 (if central venous catheter in place)
Population: None of the patients had a central venous line, so no samples were obtained for analysis.
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Central Venous Pressure (CVP).
Description: CVP
Time Frame: Change in CVP from Day 0 to 3 (if central venous catheter in place)
Population: A central venous line was not in place for the subjects so measurements could not be obtained
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Mean Arterial Pressure (MAP).
Description: MAP
Time Frame: Change in MAP from Day 0 to day 7
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 10 | 4
mm Hg | -9.96 (15.5) | 8.18 (13.1)
Statistical Analysis 1: Comparison: Treprostinil Inhalation Solution vs Placebo; Test type: Superiority; p = 0.567, Mixed Models Analysis; Measurement of MAP were evaluated from baseline to end of treatment

9. Secondary Outcome: All-cause Mortality
Description: All-cause mortality
Time Frame: 0-28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 10 | 4
Participants | 4 | 0
Statistical Analysis 1: Comparison: Treprostinil Inhalation Solution vs Placebo; Test type: Superiority; p = 0.2507, Fisher Exact — The threshold for statistical significance was 0.05

10. Secondary Outcome: Number of Subjects Requiring Intubation and Mechanical Ventilation
Description: Intubation / Mechanical Ventilation
Time Frame: 0-28 days
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 10 | 4
Participants | 4 | 0

11. Secondary Outcome: Number of Deaths During Hospitalization
Description: Hospital Mortality
Time Frame: Deaths during hospitalization (up to 3 months)
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 10 | 4
Participants | 3 | 0
Statistical Analysis 1: Comparison: Treprostinil Inhalation Solution; Test type: Superiority; p = 0.5055, Fisher Exact

12. Secondary Outcome: Peak Plasma Concentration Determined 15 Min After Inhalation and Trough Determined 4 Hours Following the Drug/Placebo Administration
Description: Treprostinil Plasma Concentration
Time Frame: Day 3
Population: Only 3 plasma pharmacokinetic samples were collected from subjects treated with Treprostinil and therefore no measurements of plasma Treprostinil were made.
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Days From Study Enrollment Until Mechanical Ventilation is Required
Description: Time to intubation and mechanical ventilation
Time Frame: Day 0 to day 28
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treprostinil Inhalation Solution | Placebo
Number analyzed (Participants) | 10 | 4
days | 2.8 (2.2) | 0 (0)

ADVERSE EVENTS:
Time Frame: From time of enrollment until end of follow-up, approximately 28 days.
Arm/Group | Treprostinil Inhalation Solution | Placebo
All-Cause Mortality (participants affected / at risk) | 4/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 4/10 | 0/4
Other Adverse Events (participants affected / at risk) | 6/10 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil Inhalation Solution (N=10) | Placebo (N=4)
Death (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0
septic shock (Infections and infestations) | 1 (1) | 0 (0)
Transfusion Reaction (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil Inhalation Solution (N=10) | Placebo (N=4)
Nausea/Emesis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Cholelithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Metapneumovirus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediatinum/Bilateral pneumothoraces (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Retro-peritoneal hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Sleep Interference (General disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Hypernatremia (Renal and urinary disorders) | 1 (1) | 1 (1)
Transfusion Reaction (Immune system disorders) | 1 (1) | 0 (0)
GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Hyponatremia (Renal and urinary disorders) | 1 (2) | 0 (0)
Elevated Transaminase (Gastrointestinal disorders) | 1 (1) | 0 (0)
Parapneuomonic Effusion with decortication (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Delirium (Nervous system disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was stopped because of low recruitment. The limited number of subjects make it difficult to draw conclusions regarding the efficacy of Treprostinil in subjects at high risk of developing ARDS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT02370095/Prot_SAP_000.pdf